CLINICAL TRIAL: NCT05090579
Title: Nalgesic Effect of Nulbuphine-bupivacaine Combination in Ultrasound Guided Transversus Abdominis Plane Block in Patients Undergoing Major Abdominal Cancer Surgeries .
Brief Title: Comparison Between Two Different Doses of Nulbuphine _bupivacaine in TAP Block in Cancer Abdominal Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Muhammed Othman, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Q123
Record Dates: First submitted 2021-09-02; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (BN10) (Active Comparator): patients will receive an ultrasound-guided TAP block with 20 mL of 0.25% bupivacaine , 1 mL of 10 mg of nulbuphine plus 4 mL of normal saline to reach 25 mL as total volume on each side of the abdominal wall.
  Interventions: Procedure: Group I (BN10)
- Group II (BN20) (Active Comparator): patients will receive an ultrasound-guided TAP block with 20 mL of 0.25% bupivacaine ,2 mL of 20 mg of nulbuphine plus 3 mL of normal saline to reach 25 mL as total volume on each side of the abdominal wall.
  Interventions: Procedure: Active Comparator:Group ll (BN20)
- Group lll(B) (Active Comparator): patients will receive 20 mL of 0.25%bupivacaine plus 5 mL of normal saline to reach 25 mL as total volume on each side of the abdominal wall.
  Interventions: Procedure: Active Comparator:Group lll (B)

INTERVENTIONS:
Procedure: Group I (BN10) — patients will receive an ultrasound-guided TAP block with 20 mL of 0.25% bupivacaine, 1 mL of 10 mg of nalbuphine plus 4 mL of normal saline to reach 25 mL as total volume on each side of the abdominal wall
  Arms: Group I (BN10)
Procedure: Active Comparator:Group ll (BN20) — patients will receive an ultrasound-guided TAP block with 20 mL of 0.25% bupivacaine, 2 mL of 20 mg of nalbuphine plus 3 mL of normal saline to reach 25 mL as total volume on each side of the abdominal wall
  Arms: Group II (BN20)
Procedure: Active Comparator:Group lll (B) — patients will receive 20 mL of 0.25%bupivacaine plus 5 mL of normal saline to reach 25 mL as total volume on each side of the abdominal wall
  Arms: Group lll(B)

SUMMARY:
To compare the analgesic effect of two different doses of nulbuphine (10 mg and 20 mg) added to bupivacaine in bilateral subcostal single injection in ultrasound-guided TAP block for abdominal surgeries.

DETAILED DESCRIPTION:
The ultrasound-guided TAP block will be performed before the induction of general anesthesia. Upon arrival at the operating room, the patients will be place in the supine position and an 18-gauge intravenous (IV) cannula will be inserted for IV fluid and drug administration. Basic monitoring probes (electrocardiography, non-invasive blood pressure, oxygen saturation, and temperature) will be applied, and their baseline vital signs will be recorded. Lactated Ringer's solution 10mL/ kg will be infused intravenously over 10 minutes before the initiation of the TAP block.

The TAP block will be performed with the use of ultrasound, under complete aseptic technique. A broadband linear array probe will be used with an imaging depth of 4 - 6 cm. The ultrasound probe will be placed transversely to the abdomen (horizontal plane) in the midaxillary line between the costal margin and the iliac crest. Three muscle layers are clearly seen in the image. The needle (22-gauge x 80 mm SonoPlex stim cannula, Pajunk®, Geisingen, Germany) will be inserted in a sagittal plane approximately 3 - 4 cm medial to the ultrasound probe. The point of needle insertion will be closer to the probe. For optimal imaging of the needle, it will be held parallel to the long axis of the probe (in-line view). The needle tip will be directed into the plane below the internal oblique and above the transversus abdominis muscle. A small volume of local anesthetic (2 mL) was seen to open the plane between the 2 muscles and was followed by insertion of the full dose of local anesthetic. If the 2 mL dose appears to be within the muscle rather than between them, then needle adjustment will be required. The local anesthetic injected appeared hypoechoic (black compared to the muscle layers) on ultrasound image.

The TAP block will be performed with the use of ultrasound under complete aseptic technique. A broadband linear array probe will be used with an imaging depth of 4 - 6 cm using a 22-gauge × 80 mm SonoPlex stim cannula (Pajunk®, Geisingen, Germany). Twenty minutes after the TAP block, the extent of sensory blockade will be evaluated by using the pin prick test (0 = no block, 1 = hyposthesia, and 2 = anesthesia) by another blinded attending anesthetist. Any patients with a failed block will be excluded from the studied groups.

Anesthetic Technique:

The anesthetic technique will be standardized in the 3 groups. No preoperative analgesics will be given. After a successful TAP block, ?? general anesthesia will be induced intravenously (propofol 1 - 2 mg/kg, lidocaine 1.5 mg/ kg) and fentanyl 1 μg/kg. Endotracheal intubation will be facilitated by neuromuscular blockade with cisatracurium 0.3 mg/kg. Anesthesia and muscle relaxation will be maintained with isoflurane in an air/oxygen mixture and cisatracurium 0.15 mg/kg. The patients will be mechanically ventilated in parameters that maintain the end-tidal CO2 (ETCO2) between 33 and 36 mmHg. The patients' heart rate, oxygen saturation, ETCO2, and systolic and diastolic blood pressures will be measured and recorded. Hypotension will be defined as a 15% decrease in systolic blood pressure from the base line, bradycardia as a heart rate slower than 50 beats per minute, and hypoxia as an oxygen saturation less than 90%. Hypotension will be treated with intravenous boluses of ephedrine 0.1 mg/kg, repeated as required. Bradycardia will be treated with intravenous atropine 0.01 mg/kg.

At the end of surgery, muscle relaxation will be reversed by neostigmine 50 μg/kg and atropine 10 μg/ kg. The patients will be extubated and transferred to the post-anesthesia care unit (PACU), where they will be monitored for vital signs (heart rate, non-invasive blood pressure, respiratory rate, and O2 saturation) immediately postoperatively and at 2, 4, 6, 12, 18, and 24 hours postoperatively.

The severity of pain and the presence of nausea, vomiting, and respiratory depression will be assessed postoperatively at 0, 2, 4, 6, 12, 18 and 24 hours. The severity of pain will be assessed using a 10 cm VAS at rest and coughing (0 = no pain and 10 = worst imaginable pain). Repiratory function : FVC, FEV and FEV1 /FVC ratio will be recorded postoperatively and 6,12,&24 hr. Postoperatively. If a patient's VAS score was ≥ 3, morphine will be administered intravenously by a dose of 0.05 mg/kg at 15minute intervals until complete pain relief will be achieved. Morphine administration will be ceased when the VAS score at rest and coughing was < 3 on assessment or when over-sedation or respiratory depression will occur (a respiratory rate of < 10 bpm). Rescue antiemetic will be given in the form of ???metoclopramide 10 mg (Zofran 4mg) IV when patients complained of nausea or vomiting.???? (Our primary outcome measure will be total morphine consumption in the first 24 hours postoperatively; our secondary outcome measures will be the postoperative VAS scores, the time of the first request of rescue analgesia (calculated from the time of the TAP block application), spirometry lung function testing and the incidence of postoperative side effects)

ELIGIBILITY:
Inclusion Criteria:-

* ASA classification I-ll,
* Aged >18 years,
* weight 50-85 kg,
* Patients who will undergo abdominal cancer surgery.

Exclusion Criteria:-

* Patient's refusal,
* patients with a history of allergies to studied drugs,
* Patients with coagulation disorders,
* Patients with opioid dependence,
* Patients with morbid obesity (body mass index more than 40 kg/m2),
* Patients with sepsis,
* patients with psychiatric illnesses that will interfere with the perception and assessment of pain .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
time of request of first analgesia | Time Frame: 24 hours post-operatively ]
  VAS (Visual Analogue Scale, 0-100 mm; where 0 = no pain, and 100 = worst imaginable pain) will be assessed, at rest, per hour for 24 hours post operatively. Moreover, VAS will also be assessed at 12 and 24 hours post-operatively while abducting the ipsilateral arm. If the patient experiences a pain of > 3, IV morphine will be given at a dose of 2.5-5 mg per dose, with a maximum dose of 10 mg, aiming for a pain score of ≤ 3. Time which will pass until the request of first analgesia shall be determined for each group and compared.

SECONDARY OUTCOMES:
total morphine consumption in the first 24 hours postoperatively | Time Frame: 24 hours post-operatively ]
  If a patient's VAS score was ≥ 3, morphine will be administered intravenously by a dose of 0.05 mg/kg at 15 minute intervals until complete pain relief will be achieved. Morphine administration will be ceased when the VAS score at rest and coughing was < 3 on assessment or when over-sedation or respiratory depression will occur (a respiratory rate of < 10 bpm). Rescue antiemetic will be given in the form of ondasteron 4 mg IV when patients complained of nausea or vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Rania M. Abdel -Emam, Study Director — South Egypt cancer Institute, Assuit university hospitals; Shreen M. Muhammed, A.professor, Study Director — South Egypt cancer Institute, Assuit university hospitals; Eman A. Ismail, Study Chair — Assiut University hospitals
Locations (1):
- Amira Muhammed Othman, Asyut, Egypt